CLINICAL TRIAL: NCT06113900
Title: Assessment of Safety and Efficacy of Sodium Glucose Co-transporter 2 Inhibitors Among Lupus Nephritis Patients
Brief Title: Assessment of Safety and Efficacy of SGLT2is Among LN Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Mohamed Ahmed Waly, Head of Nephrology Department, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SGLT2I among LN patients
Record Dates: First submitted 2023-09-20; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — dapagliflozin; empagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug as Dapagliflozin 10 mg orally for 6 months is given (Experimental): 25 lupus nephritis patients will receive SGLT2is as dapagliflozin 10mg beside there usual treatment of lupus for 6 months
  Interventions: Drug: Dapagliflozin 10mg Tab orally once daily
- On there conventional lupus nephritis treatment (No Intervention): 25 lupus nephritis patients didn't receive SGLT2i and continue on their conventional lupus nephritis treatment

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab orally once daily — Sodium glucose co-transporter 2 inhibitors
  Other Names: Empagliflozin 10 mg tab orally once daily
  Arms: Drug as Dapagliflozin 10 mg orally for 6 months is given

SUMMARY:
The aim of this study is to assess the safety and efficacy of SGLT2is among LN patients.

DETAILED DESCRIPTION:
SLE is a chronic debilitating autoimmune disorder that involves multiple organ systems either simultaneously or sequentially with relapsing and remitting course. The word 'Lupus' is a Latin term which means wolf.

Lupus nephritis (LN) is one of the common complications in patients with SLE and influences overall outcome of these patients. About two-thirds of patients with SLE have renal disease at some stage which is a leading cause of mortality in these patients.

Manifestations of LN vary from asymptomatic urinary abnormalities to rapidly progressive crescentic glomerulonephritis to end-stage renal disease (ESRD).

Recently, metabolic modulation approach has become a hot spot in the management of SLE. Increased glucose metabolism in immune cells has been reported in patients with SLE.

Repurposing metformin, an old anti diabetic drug, has the potential to reduce the risk of lupus flare in randomized controlled trials. A recent crossover study implied that peroxisome proliferator-activated receptor-gamma agonists might decrease cardiovascular risk in patients with SLE.

Dapagliflozin, SGLT2i, is a new therapy for type 2 diabetes. The Dapagliflozin mode of action is to reduce glucose reabsorption in the epithelial cells of the proximal renal tubule of the kidney, which results in decreased blood glucose and glycated hemoglobin levels.

Strikingly, four cardiovascular outcome trials demonstrated that treatment with SGLT2is (empagliflozin, canagliflozin and dapagliflozin) in patients with type 2 diabetes had prominent effects on slowing the decline rate of eGFR and decreasing albuminuria, as well as a significant reduction in cardiovascular events.

Furthermore, the nephroprotective efficacy of SGLT2is was extended to non-diabetic CKD, such as IgA nephropathy.

The net gain of SGLT2 inhibition is to reduce renal workload and to modulate weight loss and blood pressure.

The paradigm for CKD and congestive heart failure management has been shifted accordingly

Interestingly, all researchers have reported that SGLT2is could block lipopolysaccharide-induced and NLRP3-mediated inflammatory responses and regulate macrophage polarization via interplay with mammalian target of rapamycin (mTOR) and AMP-activated protein kinase pathway thereby, SGLT2is might further contribute to reducing inflammation, modulating endothelial dysfunction and decelerating atherosclerosis which are all relevant to the pathophysiology of SLE.

Here, the investigators initiated this study aiming to assess the safety and efficacy of dapagliflozin among patients with LN.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 year.
* Patients with confirmed SLE according to EULAR/ACR classification criteria.
* Patients with LN ( persistent proteinuria > 2 gm per day or greater than 3+ by dipstick, and/or cellular casts including red cell, hemoglobin, granular, tubular or mixed & "active urinary sediment" (>5 RBC/hpf, >5 WBC/hpf in the absence of infection, or cellular casts limited to RBC or WBC casts )
* Patient with e GFR > 25 ml/min/1.73m2 by CKD-EPI equation.

Exclusion Criteria:

* Patients with an allergy or intolerance to Dapagliflozin or any prior SGLT2i exposure within 1 month before screening.
* Medical history of chronic disease (Severe respiratory distress, gastrointestinal tract lesions & chronic liver disease)
* Patients with recurrent genitourinary infections.
* Patient with proteinuria < 2gm.
* Patient who show response to immune therapy in proteinuria reduction > 50%.
* Patient with Lupus in induction phase.
* Patient on steroids > 30 mg daily dose.
* Patients with diabetes mellitus.
* Patients with severe infection requiring antibiotics within 1 month before screening.
* Patients with malignant diseases.
* Pregnant or breast-feeding women.
* Patients with eGFR < 25 ml/min/1.73m2 or undergoing dialysis therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Renal Function Tests: | 6 months
  1. Measurement of serum urea level in mg/dl at 3 month's interval, that is, at 0, 3 and 6 months.
  2. Measurement of serum creatinine level in mg/dl at 3 month's interval, that is, at 0, 3 and 6 months.
  3. Measurement of serum uric acid level in mg/dl at 3 month's interval, that is, at 0, 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Howaida Al-Shennawi, Professor, Principal Investigator — Professor of internal medicine and Nephrology; Cherry Kamel, Professor, Study Director — Professor of internal medicine and Nephrology
Locations (1):
- Ain Shams University, Alexandria, Egypt

REFERENCES:
- [Background] Abdollahi E, Keyhanfar F, Delbandi AA, Falak R, Hajimiresmaiel SJ, Shafiei M. Dapagliflozin exerts anti-inflammatory effects via inhibition of LPS-induced TLR-4 overexpression and NF-kappaB activation in human endothelial cells and differentiated macrophages. Eur J Pharmacol. 2022 Mar 5;918:174715. doi: 10.1016/j.ejphar.2021.174715. Epub 2022 Jan 11. PMID 35026193
- [Background] Braunwald E. Gliflozins in the Management of Cardiovascular Disease. N Engl J Med. 2022 May 26;386(21):2024-2034. doi: 10.1056/NEJMra2115011. No abstract available. PMID 35613023
- [Background] Gounden V, Bhatt H, Jialal I. Renal Function Tests. 2024 Jul 27. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK507821/ PMID 29939598
- [Background] Ma Y, Zhao Q, Peng H, Nalisa DL, Shan P, Jiang H. SGLT2i in Patients with Type 1 Diabetes: Benefits, Risks, and Preventive Strategies. Front Biosci (Landmark Ed). 2023 May 22;28(5):98. doi: 10.31083/j.fbl2805098. PMID 37258468
- [Background] Parodis I, Gomez A, Lindblom J, Chow JW, Sjowall C, Sciascia S, Gatto M. B Cell Kinetics upon Therapy Commencement for Active Extrarenal Systemic Lupus Erythematosus in Relation to Development of Renal Flares: Results from Three Phase III Clinical Trials of Belimumab. Int J Mol Sci. 2022 Nov 11;23(22):13941. doi: 10.3390/ijms232213941. PMID 36430417
- [Background] Sada K, Kurita N, Noma H, Matsuki T, Quasny H, Levy RA, Jones-Leone AR, Gairy K, Yajima N. MOONLIGHT study: the design of a comparative study of the effectiveness of belimumab in patients with a history of lupus nephritis from the post-Marketed effectiveness of belimumab cOhOrt and JapaN Lupus NatIonwide reGistry (LUNA) coHorT. Lupus Sci Med. 2022 Sep;9(1):e000746. doi: 10.1136/lupus-2022-000746. PMID 37017254
- [Derived] Desai SB, Ahdoot R, Malik F, Obert M, Hanna R. New guidelines and therapeutic updates for the management of lupus nephritis. Curr Opin Nephrol Hypertens. 2024 May 1;33(3):344-353. doi: 10.1097/MNH.0000000000000969. Epub 2024 Feb 9. PMID 38334499